CLINICAL TRIAL: NCT00914108
Title: Family-Centered Neuropsychoeducational In-NICU Intervention for Preterm Infants With Severe Intrauterine Growth Retardation and for Their Families
Brief Title: Severe Intrauterine Growth Retardation: Developmental Newborn Intensive Care Unit (NICU) Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Heidelise Als, PhD, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: X03-10-072R
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Intrauterine Growth Retardation; Prematurity
Keywords: Preterm Infants; Developmental Care; NIDCAP; Intrauterine Growth Restriction; APIB; EEG; Neurobehavior
MeSH Terms: conditions — Fetal Growth Retardation; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Newborn Individualized Developmental Care — The developmental care model aims to create a relationship-based developmentally supportive care environment for the preterm infant and family. The theory proposes that care implementation that takes into account infants' thresholds of disorganization is most supportive of long term outcome. Specifically, the intervention consisted of weekly neurobehavioral observations and reports of the experimental group infants' behavior with suggestions for parents and staff in ways to support each infant's development. The developmental specialists observed each infant's behavior throughout hospitalization and to 2 weeks corrected age and formulated descriptive neurobehavioral reports with suggestions to structure caregiving procedures adapted to the infant's sleep/wake cycle and in support of the infant's well-regulated behavioral balance. Parents were supported to care for their infant, encouraged to nurse and hold their infant skin-to-skin, and to cradle them during stressful procedures.
  Other Names: NIDCAP

SUMMARY:
The purpose of the study is to learn more about the development of small for gestational age (SGA) preterm infants and whether focusing on the infant's behavior has a positive effect on outcome. The study hypotheses state: 1) High risk severely SGA preterm infants will profit from detailed neuropsychological assessment, psychoeducational recommendations and practical guidance for caregiving, as well as formal educational and emotional support for the family and the professional care team. 2) Neuropsychological education and guidance for community-based early intervention providers caring for SGA preterm infants after their discharge is effective in promoting improved outcome.

DETAILED DESCRIPTION:
The preterm infant who is not only born early but also did not grow well in the womb is at double jeopardy for developmental disabilities. The literature indicates that the fetus who has not gained weight properly nor is showing expected head growth in the womb [symmetrical intrauterine growth retardation (IUGR) or small for gestational age (SGA) status] will not only require significantly longer stays in the newborn intensive care unit (NICU) and grow more poorly than the appropriately grown prematurely born infant, but will also show significant disabilities later on in terms of fine and gross motor skills, cognitive function activity, language abilities, abstract reasoning, concentration, attention, mood and temperament. IUGR exerts an independent adverse effect on the developmental outcome of preterm infants.

Given the importance of the last 4 months of gestation and the first 2 years post term for brain growth and development, and given the relationship between cerebral development and behavior which is a two-way street and a dynamic feedback system, the particular vulnerability of SGA children to environmental factors indicates that there are grounds for the hypothesis that appropriate support and intervention for severely SGA preterm infants and their families might ameliorate dysfunction.

The general purpose of the proposed project is to develop and test a model of ameliorative neuropsychoeducational intervention in the NICU in support of the developmental outcome of severely SGA preterm infants and their families. The specific hypotheses to be tested are as follows:

1. High risk severely SGA preterm infants cared for in the NICU with the support of a neuropsychoeducational model of intervention will show:

   1. At 2 weeks post term, more well-regulated autonomic, motor, state organizational and attentional functioning
   2. At 9 and 24 months post term:

      * More well-regulated autonomic and visceral functioning with less colic and improved eating patterns and weight gain
      * More well-regulated motor system performance
      * More well-regulated state organization, including sleep and awake organization
      * More well-regulated cognitive and attentional functioning in various domains, including visual-motor integration, spatial planning, attentional planning, expressive and receptive language function, abstract verbal reasoning, short term memory and continuous performance regulation
      * More well-regulated executive function capacities
      * More well-regulated affective emotional functioning
2. Parents whose infants receive the support of a neuropsychoeducational model of care will show:

   1. At 2 weeks, 9 and 24 months post term, enhanced appreciation of their infant as an individual
   2. At 9 and 24 months post term, more sensitively attuned input in support of their child's functioning, more competent parenting strategies, and a greater sense of effectiveness in parenting the child.

The population will consist of severely small for gestational age preterm infants admitted to the NICU and randomly assigned to a control and experimental group.

Effectiveness of the experimental treatment for the experimental group will be tested at three systematic outcome points in various domains. The domains assessed include (1) medical outcome; (2) neurobehavioral outcome; (3) neuroelectrophysiological outcome; and (4) family outcome. The outcome points for infant and family are 2 weeks, 9 and 24 months after expected due date.

The study is expected to demonstrate intervention effectiveness in improving IUGR preterm infants' neurodevelopment. It is anticipated that the results will set the stage for a model of caregiving and intervention that lives up to the mandate that every child is entitled to an environment, care and education appropriate to his or her specific needs. The model can then be used in other nurseries to provide improved outcome for preterm populations.

ELIGIBILITY:
Inclusion Criteria:

* Inborn at the Brigham and Women's Hospital
* Gestational age < 36 weeks
* Birthweight < 5th percentile
* Head circumference at birth < 5th percentile

Exclusion Criteria:

* Presence of major chromosomal or congenital anomalies (Down's, Turner's, Klinefelter's Syndrome, etc.)
* Presence of major congenital infections (HIV, TORCH)
* Presence of significant prenatal focal brain lesions (intrauterine infarcts; cystic changes, etc.)
* Presence of major maternal illness (uncontrolled diabetes, active seizure disorder requiring medication during pregnancy, renal transplant), mental and/or emotional impairment (including heroin addiction and documented alcoholism)

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 1996-10; Primary Completion 2000-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Evidence of improved neurodevelopmental and neurophysiological outcome as assessed with: Assessment of Preterm Infants' Behavior (APIB) and electrophysiological (EEG) assessment | At 2 weeks , 9 months and 24 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Heidelise Als, PhD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts

REFERENCES:
- [Derived] McAnulty G, Duffy FH, Kosta S, Weisenfeld NI, Warfield SK, Butler SC, Alidoost M, Bernstein JH, Robertson R, Zurakowski D, Als H. School-age effects of the newborn individualized developmental care and assessment program for preterm infants with intrauterine growth restriction: preliminary findings. BMC Pediatr. 2013 Feb 19;13:25. doi: 10.1186/1471-2431-13-25. PMID 23421857
- [Derived] Als H, Duffy FH, McAnulty G, Butler SC, Lightbody L, Kosta S, Weisenfeld NI, Robertson R, Parad RB, Ringer SA, Blickman JG, Zurakowski D, Warfield SK. NIDCAP improves brain function and structure in preterm infants with severe intrauterine growth restriction. J Perinatol. 2012 Oct;32(10):797-803. doi: 10.1038/jp.2011.201. Epub 2012 Feb 2. PMID 22301525
- [Derived] Als H, Duffy FH, McAnulty GB, Fischer CB, Kosta S, Butler SC, Parad RB, Blickman JG, Zurakowski D, Ringer SA. Is the Newborn Individualized Developmental Care and Assessment Program (NIDCAP) effective for preterm infants with intrauterine growth restriction? J Perinatol. 2011 Feb;31(2):130-6. doi: 10.1038/jp.2010.81. Epub 2010 Jul 22. PMID 20651694